CLINICAL TRIAL: NCT03463473
Title: First-in-human, Open-label, Phase 1 Dose-Escalation Study of MSB2311, A Humanized Anti-PD-L1 Monoclonal Antibody in Subjects With Advanced Solid Tumors
Brief Title: A Phase I Study of MSB2311 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MSB2311-CSP-001
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2019-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Dose escalation : 3mg/kg Q3W, 10 mg/kg Q3W, 20 mg/kg Q3W, 10 mg/kg Q2W
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 3 mg/kg (Q3W) MSB2311 Injection (Experimental): MSB2311 will be administered as an IV infusion once every 3 weeks (Q3W) starting at 3 mg/kg.
  Interventions: Drug: 3 mg/kg Q3W MSB2311 Injection
- 10 mg/kg (Q3W) MSB2311 Injection (Experimental): MSB2311 will be administered as an IV infusion once every 3 weeks (Q3W) starting at 10 mg/kg.
  Interventions: Drug: 10 mg/kg Q3W MSB2311 Injection
- 20 mg/kg (Q3W) MSB2311 Injection (Experimental): MSB2311 will be administered as an IV infusion once every 3 weeks (Q3W) starting at 20 mg/kg.
  Interventions: Drug: 20 mg/kg Q3W MSB2311 Injection
- 10 mg/kg (Q2W) MSB2311 Injection (Experimental): MSB2311 will be administered as an IV infusion once every 2weeks (Q2W) starting at 10 mg/kg.
  Interventions: Drug: 10 mg/kg Q2W MSB2311 Injection

INTERVENTIONS:
Drug: 3 mg/kg Q3W MSB2311 Injection — An intravenous infusion with concentration from 3 mg/kg (Q3W)
  Other Names: 3 mg/kg Q3W MSB2311
  Arms: 3 mg/kg (Q3W) MSB2311 Injection
Drug: 10 mg/kg Q3W MSB2311 Injection — An intravenous infusion with concentration from 10 mg/kg (Q3W)
  Other Names: 10 mg/kg Q3W MSB2311
  Arms: 10 mg/kg (Q3W) MSB2311 Injection
Drug: 20 mg/kg Q3W MSB2311 Injection — An intravenous infusion with concentration from 20 mg/kg (Q3W)
  Other Names: 20 mg/kg Q3W MSB2311
  Arms: 20 mg/kg (Q3W) MSB2311 Injection
Drug: 10 mg/kg Q2W MSB2311 Injection — An intravenous infusion with concentration from 10 mg/kg (Q2W)
  Other Names: 10 mg/kg Q2W MSB2311
  Arms: 10 mg/kg (Q2W) MSB2311 Injection

SUMMARY:
This is a phase I study to determine the safety and toxicity, PK/PD, immunogenicity, biomarkers, anti-tumor activity and establish a preliminary recommended Phase 2 dose (RP2D) in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), open-label, Phase 1 dose-Escalation Study of MSB2311, a humanized anti-PD-L1 monoclonal antibody, in subjects with advanced solid tumors. Qualified subjects will be enrolled to receive their assigned dose regimen of MSB2311 until disease progression or intolerable toxicity, withdrawal of consent, or end of study, whichever occurs first. The maximum treatment duration is 2 years. During the study, subjects will be evaluated for safety and toxicity, PK/PD, immunogenicity, biomarkers, and anti-tumor activity of MSB2311.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign the ICF.
* Male or female subject ≥ 18 years.
* Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumors that are refractory to standard therapy, or for which no standard therapy exists.
* Subject has measurable disease per RECIST v1.1.
* ECOG Performance Status 0 to 1
* Subjects with life expectancy of ≥ 3 month
* No herbal/alternative medications prior to the first dose
* Must have adequate hematological, hepatic and renal function as defined in the protocol.
* Prior anti-tumor therapies of different kinds must have stopped before the first dose as defined by protocol
* Effective contraception for both male and female subjects if the risk of conception exists

Exclusion Criteria:

* Pregnant or nursing females.
* Any remaining AEs > grade 1 from prior anti-tumor treatment as per CTCAE v4. 03, with exception of the residual hair loss;
* Received a biologic G-CSF, GM-CSF or erythropoietin within 14 days prior to the first dose of study drug;
* Subjects who had prior treatment with an anti-PD-L1 product
* History of documented autoimmune disease except for autoimmune hypothyroidism and well-controlled Type 1 diabetes mellitus.
* W/o autoimmune condition requiring systemic treatment with immunosuppressive medications within 14 days before the planned first dose of study drug.
* Primacy central nervous system (CNS) malignancy or symptomatic CNS metastases are not allowed, with exceptions defined in protocol.
* Major surgery within the 28-days from the screening
* Subjects with idiopathic pulmonary fibrosis or unresolved active or chronic inflammatory pulmonary disease are excluded.
* History of human immunodeficiency virus (HIV) infection, active hepatitis B or C. HBV carriers
* History of primary immunodeficiency, stem cell or organ transplant, or previous clinical diagnosis of tuberculosis disease.
* Clinically significant acute infections 4 weeks and any infection 2 weeks prior to the first dose administration.
* Known allergies, hypersensitivity, or intolerance to protein-based therapies or with a history of any significant drug allergy
* Subjects who experienced immunotherapy-related adverse events (irAE) grade ≥ 3, or who had to discontinue prior anti-PD-1 treatment due to irAEs of any grade.
* Severe or uncontrolled cardiac disease requiring treatment as defined in protocol
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, might impair the subject's benefit from the trial treatment
* Known history of hypersensitivity to any components of the MSB2311 product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MSB2311 | Up to 90 days following the last dose
  Measured by number adverse events that are related to treatment
Maximum tolerated dose or recommended phase 2 dose | Up to 90 days following the last dose
  Measured by number of subjects experiencing DLT in each escalation cohort

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) for MSB2311 | Up to 30 days following the last dose
Peak Plasma concentration (Cmax)for MSB2311 | Up to 30 days following the last dose
  Incidence and quantity of anti-drug antibodies
Volume of plasma from which MSB2311 is completely removed per unit time (CL) | Up to 30 days following the last dose
The incidence of subjects generating anti-drug antibody | Up to 30 days following the last dose
Objective response rate (ORR) as measured by RESISTv1.1 | Up to 30 days following the last dose
Duration of response (DOR) as measured by RESISTv1.1 | Up to 30 days following the last dose
Progression-free survival (PFS) as measured by RESISTv1.1 | Up to 30 days following the last dose
Best overall response as measured by RESISTv1.1 | Up to 30 days following the last dose
Overall survival (OS) as measured by RESISTv1.1 | Up to 30 days following the last dose
Elimination half-life and apparent plasma terminal phase elimination rate constant (t1/2 ) of MSB2311 | Up to 30 days following the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Yonggang Wu, MD, Study Director — Suzhou Transcenta Therapeutics Co., Ltd.
Locations (1):
- South Texas Accelerated Research Therapeutics, San Antonio, Texas, United States